CLINICAL TRIAL: NCT01167920
Title: Virtual Hypertension Clinic (VHC) Study
Brief Title: Virtual Hypertension Clinic
Acronym: VHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-575
Record Dates: First submitted 2010-07-14; First posted 2010-07-22 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Hypertension; Home Blood Pressure Measurements; Wireless communication of measurements; Wireless communication of blood pressure measurements
MeSH Terms: conditions — Hypertension | interventions — Angiotensin-Converting Enzyme Inhibitors; Receptors, Angiotensin; Calcium Channel Blockers; Renin Inhibitors; Diuretics; Vasodilator Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Hypertension Clinic Group (Active Comparator): In the VHC group, patients will be ask to regularly measure blood pressure with the Stabil-o-Graph so that these readings are transmitted to Virtual Hypertension Clinic. The data will be reviewed weekly and the patient will receive feedback and intervention if needed at every 2 week interval to achieve blood pressure goal. Once they reach goal, the feedback will be less intense and given at four week intervals till the end of the study.
  Interventions: Other: Virtual Hypertension Clinic
- Usual Care Group (No Intervention): The Usual Care Group (UCG) patients will be told their BP is not in control and encouraged to work with their physician to improve it. There will be no further structured intervention during the rest of the study.

INTERVENTIONS:
Other: Virtual Hypertension Clinic — In the VHC group, patients will be ask to regularly measure blood pressure with the Stabil-o-Graph so that these readings are transmitted to Virtual Hypertension Clinic. The data will be reviewed weekly and the patient will receive feedback and intervention if needed at every 2 week interval to achieve blood pressure goal. Once they reach goal, the feedback will be less intense and given at four week intervals until the end of the study.
  Other Names: ACE Inhibitors; Angiotensin II Receptors; Calcium Channel Blockers; Renin Inhibitors; Diuretics; BetaBlockers; AlphaBlockers; Vasodilators
  Arms: Virtual Hypertension Clinic Group

SUMMARY:
This is a prospective, randomized controlled trial designed to determine whether blue tooth and telephone technology can be utilized to successfully relaying home blood pressure information electronically to healthcare providers so that timely and more frequent treatment interventions can be instituted to optimize and reach goal blood pressure level for an individual as compared to usual care. The primary study outcomes are improvement in systolic, diastolic, and blood pressure control and time to control blood pressure. Secondary outcomes are proportion of patients controlled to blood pressure goal at the end of the study, adherence to blood pressure monitoring and utilization of VHC model.

If this is successful and cost-effective such technology and interventions could be utilized on large scale to improve the care and proportion of hypertensive patients achieving goal blood pressure in the United States.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for renal and cardiovascular disease, and a significant contributor to adult disability. About 50 million individuals are hypertensive in the United States1. The Framingham Heart Study suggests that normotensive individuals at 55 years have a 90% lifetime risk of hypertension2. Treatment of hypertension is the leading reason for physician visits and prescription drugs in the US3. Despite increasing awareness of the risks and of complications of poorly controlled hypertension, only 58% of hypertensive patients are being treated and of these only 38% achieve blood pressure control4, 5. Sub-optimal therapy remains the most common cause for uncontrolled hypertension6. One of the major barriers to effective management of hypertension is therapeutic inertia on the part of physicians that leads to suboptimal therapy being prescribed for hypertensive patients7.

This barrier to effective hypertension treatment achieves further significance as data from several clinical trials clearly demonstrate that reduction of blood pressure by even a few millimeters of mercury can significantly decrease an individual risk for mortality from cardiovascular disease8.

Although hypertension remains the most common reason for patient visit to a physician office in the United States, the lack of patient-health care provider connectivity outside the office setting may play an important factor in the disappointing proportion of patients achieving blood pressure control in the US for the past 30 years.

Recent home blood pressure monitoring guidelines published by the American Heart Association and other professional societies have emphasized the importance of home blood pressure monitoring in the management of hypertension9. In addition, a recent study by Green et al extended this concept a step further by utilizing a web based intervention utilized by a pharmacist to control blood pressure10. Results from this study they demonstrated a significant reduction in blood pressure in the intervention group when compared to usual care (-14.2 mmHg Vs -5.3 mmHg p <0.001).

One of the potential draw backs of a web based intervention for blood pressure control could be the lack of access to internet in the general population. According to a recent USDA report, almost 40% Americans in urban areas and 60% in rural areas do not have internet access (http://arstechnica.com/tech-policy/news/2009/03/the-many-blessing-of-rural.ars ). This in essence would deprive a large number of those with hypertension from access to the web based newer models of blood pressure control as tested in the recent study by Green et al.

The Stabil-o-Graph is a validated home blood pressure device (http://www.dableducational.org/dabl_library/library2_sbpm.html#upper_arm) that relays blood pressure readings to a designated health care provider using blue tooth technology and a telephone connection

The current model of health care in the US for the management of hypertension employs direct patient-physician encounters in an office setting to control blood pressure. This existing healthcare model has failed to keep abreast with current national guidelines and consensus among experts in hypertension that promote home blood pressure monitoring and application of newer technology with the potential to seamlessly connect a patient with his health care provider with the goal of improved blood pressure control.

Our proposed study aims to address this gap in patient-healthcare provider connectivity utilizing newer technology and home blood pressure monitoring to achieve goal blood pressure foe an individual.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25-65 years with essential hypertension
* Poorly controlled Hypertension (Systolic BP 140-199 Diastolic BP 90-110 mmHg

Exclusion Criteria:

* Patient on 4 or more antihypertensive medications
* History of non compliance with medications
* If extra-large cuff cannot fit the arm
* Patient with estimated glomerular filtration of less than 30 ml/min in the past two years)
* Patients with acute glomerulonephritis
* Patient with secondary hypertension
* Patient with severe congestive heart failure (New York Heart Association Functional Classification Class III AND IV)
* Patient with cirrhosis
* Patients with terminal diseases like cancers (other than non-melanoma skin cancers)
* Excessive alcohol intake (> 7 servings/week)
* Sensitivity or contra-indications to the use of 2 or more classes of antihypertensive medications
* Women who are pregnant (self reported) or lactating
* Women on oral contraceptive pills

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
changes in home diastolic, systolic, and mean arterial blood pressure | week 0 (screening) and week 15(final week)
  BP taken at home twice a day (morning and evening) Comparison of the average of the screening week's (Week 0)home blood pressure measurements with the average of the final week's (Week 15) home blood pressure measurements for each participant. Mean arterial blood pressure measurement values obtained at Clinic Visit One and Clinic Visit Two will be compared

SECONDARY OUTCOMES:
The proportion at the end of the study of participants in each group with controlled hypertension based on average home diastolic and systolic blood pressures transmitted by Stabil-o-Graph (averaged over each 2 week interval during the study period). | Week 0(screening) and Week 15 (final)
  Comparison of the average of the screening week's (Week 0)home blood pressure measurements with the average of the final week's (Week 15) home blood pressure measurements for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Rafey, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Vasan RS, Beiser A, Seshadri S, Larson MG, Kannel WB, D'Agostino RB, Levy D. Residual lifetime risk for developing hypertension in middle-aged women and men: The Framingham Heart Study. JAMA. 2002 Feb 27;287(8):1003-10. doi: 10.1001/jama.287.8.1003. PMID 11866648
- [Background] Cherry DK, Burt CW, Woodwell DA. National Ambulatory Medical Care Survey: 2001 summary. Adv Data. 2003 Aug 11;(337):1-44. PMID 12924075
- [Background] Hajjar I, Kotchen TA. Trends in prevalence, awareness, treatment, and control of hypertension in the United States, 1988-2000. JAMA. 2003 Jul 9;290(2):199-206. doi: 10.1001/jama.290.2.199. PMID 12851274
- [Background] Ong KL, Cheung BM, Man YB, Lau CP, Lam KS. Prevalence, awareness, treatment, and control of hypertension among United States adults 1999-2004. Hypertension. 2007 Jan;49(1):69-75. doi: 10.1161/01.HYP.0000252676.46043.18. Epub 2006 Dec 11. PMID 17159087
- [Background] Yakovlevitch M, Black HR. Resistant hypertension in a tertiary care clinic. Arch Intern Med. 1991 Sep;151(9):1786-92. PMID 1888244
- [Background] Okonofua EC, Simpson KN, Jesri A, Rehman SU, Durkalski VL, Egan BM. Therapeutic inertia is an impediment to achieving the Healthy People 2010 blood pressure control goals. Hypertension. 2006 Mar;47(3):345-51. doi: 10.1161/01.HYP.0000200702.76436.4b. Epub 2006 Jan 23. PMID 16432045
- [Background] Whelton PK, He J, Appel LJ, Cutler JA, Havas S, Kotchen TA, Roccella EJ, Stout R, Vallbona C, Winston MC, Karimbakas J; National High Blood Pressure Education Program Coordinating Committee. Primary prevention of hypertension: clinical and public health advisory from The National High Blood Pressure Education Program. JAMA. 2002 Oct 16;288(15):1882-8. doi: 10.1001/jama.288.15.1882. PMID 12377087
- [Background] Pickering TG, Miller NH, Ogedegbe G, Krakoff LR, Artinian NT, Goff D; American Heart Association; American Society of Hypertension; Preventive Cardiovascular Nurses Association. Call to action on use and reimbursement for home blood pressure monitoring: a joint scientific statement from the American Heart Association, American Society Of Hypertension, and Preventive Cardiovascular Nurses Association. Hypertension. 2008 Jul;52(1):10-29. doi: 10.1161/HYPERTENSIONAHA.107.189010. Epub 2008 May 22. PMID 18497370
- [Background] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730
- [Background] Keles H, Ekici A, Ekici M, Bulcun E, Altinkaya V. Effect of chronic diseases and associated psychological distress on health-related quality of life. Intern Med J. 2007 Jan;37(1):6-11. doi: 10.1111/j.1445-5994.2006.01215.x. PMID 17199838